CLINICAL TRIAL: NCT04853550
Title: Long Term Follow-up After Ventral Hernia Repair With Strattice Mesh
Brief Title: Long-Term Follow-up After Ventral Hernia Repair With Strattice Mesh
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: AllerGen NCE Inc. (Industry)
Responsible Party: Principal Investigator, Farid Kehdy, Principal Investigator, University of Louisville
Other Study IDs: 19.0980
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Strattice Mesh — Subjects will be restrospectively identified has having undergone ventral hernia repair with Strattice mesh reinforcement. Once identified long term follow-up data will be collected.

SUMMARY:
This study will assess long-term outcomes (greater than 12 months) following ventral hernia repair with Strattice mesh reinforcement.

DETAILED DESCRIPTION:
Subjects will be retrospectively identified as having undergone operative repair of ventral hernia with Strattice mesh reinforcement during the period January 1, 2013 - November 1, 2017. Follow-up data will be collected either at a postoperative clinic visit or via telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Hernia repair with Strattice Mesh
* Age 18 or older

Exclusion Criteria:

* Under age 18
* No history of hernia repair

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone ventral hernia repair with Strattice Mesh between January 1, 2013 and November 1, 2019
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 24 Months
  Percentage of patients with recurrence at long-term (>12 months) follow-up.

SECONDARY OUTCOMES:
Quality of LIfe Questionnaire | 24 Months
  Percentage of patients with mean quality of life scores at long-term (>12 months) follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Farid Kehdy, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States